CLINICAL TRIAL: NCT03417362
Title: Delivery of Audiovisual Information on Early Medical Abortion to Women in Europe Via Digital Technology: is it Acceptable and Informative?
Brief Title: Delivery of Audiovisual Information on Early Medical Abortion
Acronym: EMAVID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NHS Lothian (Other Government)
Responsible Party: Principal Investigator, John Reynolds-Wright, Community Sexual and Reproductive Healthcare Trainee, NHS Lothian
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: AC17102; 235487 (Other: IRAS ID (UK)); 2018/0060 (Other: NHS Lothian R&D); 18/NS/0016 (Other: South East Scotland Research Ethics Committee)
Record Dates: First submitted 2018-01-24; First posted 2018-01-31 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Abortion Early; Abortion in First Trimester
Keywords: education; audiovisual; information; acceptability

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Animation (Other): Animation describing process of early medical abortion, what to expect, how to take medicines. This is prior to consultation.
  Interventions: Other: Animation
- Standard (No Intervention): Standard of Care - no animation ,standard consultation only.

INTERVENTIONS:
Other: Animation — 3 minute video describing and explaining early medical abortion, followed by questionnaire
  Arms: Animation

SUMMARY:
The majority of abortions in the United Kingdom (UK) are performed before 9 weeks (63 days) gestation using a method known as Early Medical Abortion (EMA). EMA involves an assessment visit and provision of two types of medication .

The assessment visit usually involves Ultrasound to confirm gestation, detailed personal history, safeguarding assessment and contraception planning, before arranging treatment and follow up.

The process is long and lots of information is given to women attending the service. In NHS Lothian (National Health Service, Lothian Health Board), the average appointment length for combined assessment and provision of the first part of treatment is 3 hours.

Despite how common abortion is ( 1 in 3), many women presenting for abortion care are not aware of what the procedure will involve. This may in part to the social stigma surrounding abortion and unintended pregnancy in general. This stigma can in turn result in feelings of anxiety and shame about the decision to terminate a pregnancy.

There is evidence that short videos shown to patients prior to abortion or contraception consultations can improve their ability to recall information and can make them feel more confident about the procedure.

Additionally, abortion care providers have found patients who have seen videos to be better prepared and informed and this allows consultations to progress more easily and allow greater time for discussion of contraceptive methods.

We have prepared a video approximately 3 minutes in length to provide information about EMA. It summarises the process described above using simple language and animated characters. The video has been translated into French, Portuguese and Swedish and has been adapted to reflect subtle differences in practice and law in these countries. We have partners in services in these three countries who will be conducting the trial there in accordance with this protocol and their own local ethics and clinical governance requirements.

DETAILED DESCRIPTION:
Despite abortion being a common medical procedure, many women do not have access to good quality, reliable information about it. This may stem from the stigma and shame surrounding the procedure leading to less community knowledge and experience sharing compared to other medical conditions, for example diabetes or heart disease.

Lack of knowledge and understanding about a medical procedure can cause anxiety, distress and confusion when seeing a healthcare professional, which in turn can prolong consultations.

By introducing the short video animation, we are hoping that this will give the women attending the service a basic level of knowledge about Early Medical Abortion, reduce the anxiety and worry they are experiencing by informing them, and make them feel more confident and clear during their consultations.

It has been shown in other studies that short videos in contraception and abortion consultations can have this impact, but a randomised control trial methodology has never been applied to this intervention.

In a standard initial Early Medical Abortion visit a patient will experience the following Patient Journey:

1. Arrival and registration
2. Waiting for appointment in waiting room
3. Ultrasound scan to determine gestation
4. Self taken vulvovaginal swab for Chlamydia and Gonorrhoea screening
5. Blood tests for : HIV, Syphilis, Full Blood Count, Blood Group
6. Return to the waiting room
7. Assessment consultation with healthcare professional (i.e. Specialist Nurse or Doctor)
8. Return to the waiting room
9. Treatment Consultation: to receive 'first part' of treatment i.e. Mifepristone and dates for 'second part' 24-48 hours later.
10. Leave department

In the study, the above will happen, however patients will be given a participant information sheet (at step 1 above )when they arrive in department to register. At Step 6, when the patient has returned to the waiting room, eligible patients will be approached and asked if they would like to participate and if so will be randomised to 'standard of care' or 'intervention' (i.e. the video). They will resume the Patient Journey above and will again be approached at Step 8 or Step 10 to complete the short questionnaire.

For the questionnaire: a single researcher will record, on a standard proforma, what information the subject had taken from the consultation and its accuracy, and the overall acceptability of the consultation using a Likert scale to quantify descriptors such as 'helpful', 'informative', 'understandable', 'impersonal', 'sympathetic' 'unsympathetic' etc.

The number of women declining to participate in the study would be recorded .

ELIGIBILITY:
Inclusion Criteria:

1. Female
2. Pregnant
3. Presenting for Termination of Pregnancy
4. Aged 16 years or over
5. Able to understand English (the video is in English, and whilst translations are available, their content has been altered to reflect abortion laws in other countries)
6. Gestation of 9 weeks (63 days) or less on ultrasound scan
7. Able to provide consent

Exclusion Criteria:

1. Non pregnant
2. Pregnancy of Unknown Location
3. Uncertain of decision or wishing to continue pregnancy
4. 15 years old or younger
5. Unable to understand English
6. Gestation 9 weeks and 1 day (64 days) or greater on ultrasound scan.
7. Unable to provide consent

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2019-03-12 (Actual); Study Completion 2019-03-12 (Actual)

PRIMARY OUTCOMES:
Is the recall of key information about EMA similar after watching the video compared to following face to face contact with a clinician? | Immediately during questionnaire
  The patient will be asked to recall any facts that they learned from watching the video/from the consultation and this will be compared to a list held by the researcher. A numerical score for points recalled will be generated for each patient.

SECONDARY OUTCOMES:
What place/ role do women who watch the video feel that it has (if any)? | Immediately during questionnaire
  Open ended questions in the questionnaire to ask participants their thoughts on video and when/where it could be viewed in relation to their treatment. The participant can select an answer from a list of options or volunteer their own.
Do women find it acceptable to receive information about Early Medical Abortion (EMA) via an animated video? | Immediately during questionnaire
  Likert Scale completed with researcher around a series of different statements relating to their acceptability of the video. Positive responses will be grouped and an overall result of 'acceptable' or 'not acceptable' will be assigned per case.

CONTACTS AND LOCATIONS:
Overall Officials: Sharon T Cameron, FRCOG, Study Director — NHS Lothian
Locations (3):
- Assistance Publique Hopitaux de Paris, Paris, France
- Karolinska University Hospital, Stockholm, Sweden
- Chalmers Centre for Sexual and Reproductive Health, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Only anonymised responses to questionnaire will be shared between sites.

REFERENCES:
- [Background] Michie L, Cameron ST, Glasier A, Johnstone A. Giving information about the contraceptive implant using a DVD: is it acceptable and informative? A pilot randomised study. J Fam Plann Reprod Health Care. 2016 Jul;42(3):194-200. doi: 10.1136/jfprhc-2015-101186. Epub 2015 Aug 6. PMID 26250853
- [Background] Powell-Jackson R, Glasier A, Cameron ST. Benefits of using a digital video disk for providing information about abortion to women requesting termination of pregnancy. Contraception. 2010 Jun;81(6):537-41. doi: 10.1016/j.contraception.2010.01.015. Epub 2010 Feb 19. PMID 20472123
- [Derived] Reynolds-Wright JJ, Belleuvre F, Daberius A, Faucher P, Gemzell-Danielsson K, Cameron ST. Information on early medical abortion for women using an audiovisual animation vs face-to-face consultation: A consortium randomized and quasi-randomized trial. Acta Obstet Gynecol Scand. 2020 Dec;99(12):1611-1617. doi: 10.1111/aogs.13944. Epub 2020 Jul 12. PMID 32573767
- See also: NHS Scotland Information and Statistics Division. Sexual Health. Abortion activity in 2016 — https://www.isdscotland.org/Health-Topics/Sexual-Health/Publications/2017-05-30/2017-05-30-Terminations-2016-Report.pdf